CLINICAL TRIAL: NCT03828058
Title: A 12 Month Single-center, Open Label, Randomized, Comparative Study to Evaluate Envarsus XL Steroid-free Rabbit Anti-thymocyte Globulin Induction on Renal Function and Health-related Quality of Life Following Liver Transplantation
Brief Title: Envarsus XL Immunosuppression Following Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Methodist Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-05876-FB
Record Dates: First submitted 2018-12-11; First posted 2019-02-04 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Recipients of Liver Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: The study will be a prospective, randomized, open label study comparing Envarsus XR with twice daily prograf.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Envarsus XR (Experimental): Envarsus XR orally administered Daily
  Interventions: Drug: Envarsus XR
- Prograf (Active Comparator): Prograf PO administered twice daily Generic Name: tacrolimus
  Dosage of prograf will be determined by trough levels and adjusted accordingly
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Envarsus XR — Envarsus XR to be administered orally, once a day. Dosage will be adjusted as determined by trough blood levels.
  Other Names: ENVARSUS XR 0.75Mg Extended-Release Tablet; ENVARSUS XR 1Mg Extended-Release Tablet; ENVARSUS XR 4Mg Extended-Release Tablet
  Arms: Envarsus XR
Drug: Prograf — Prograf 2 mg BID to be administered orally, twice a day. Dosage will be adjusted as determined by trough blood levels.
  Other Names: Tacrolimus
  Arms: Prograf

SUMMARY:
The standard immunosuppressive regimen for liver transplantation includes twice daily tacrolimus (Prograf). In other transplantation models, there are potential benefits to extended release formulations as lower peak concentrations are thought to have lower rates of nephrotoxicity. Additionally, compliance with once daily medications is felt to be easier than twice daily medications. Our aim is to look at our prospective liver transplant group and see if once daily tacrolimus (Envarsus XR) results in improved renal function as well as improved health care quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or older
4. Recipients of a first-time liver transplant
5. Serum Creatinine level less than 2.0 on Post-Operative Day 3-7
6. Ability to take oral medication and be willing to adhere to the assigned immunosuppression regimen
7. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

1. Any prior use of tacrolimus or cyclosporine
2. Recipients of prior organ transplant
3. Need for hemodialysis in the week preceding or following liver transplantation
4. Recipients of living donor liver or split deceased donor liver allografts
5. Recipients of combined liver/kidney transplants
6. Pregnancy or lactation
7. Recipients of ABO incompatible liver allografts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) over the first year after liver transplant | 3, 6, and 12 months post-transplant
  We will be assessing differences in renal function based on calculated eGFR by MDRD6 equation.

SECONDARY OUTCOMES:
Quality of Life Assessment | 3, 6, and 12 months post-transplant
  We will be using the RAND Short Form 36 (SF36) healthcare survey to assess patient reported quality of life across a broad spectrum ranging from physical health and function to emotional well being. Each sub scale score ranges from 0 (worse) to 100 (best).

CONTACTS AND LOCATIONS:
Overall Officials: James Eason, MD, Study Director — The University of Tennessee Health Science Center, Department of Transplant
Locations (1):
- Methodist Healthcare, University Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kadam P, Bhalerao S. Sample size calculation. Int J Ayurveda Res. 2010 Jan;1(1):55-7. doi: 10.4103/0974-7788.59946. No abstract available. PMID 20532100
- [Result] Abdelmalek MF, Humar A, Stickel F, Andreone P, Pascher A, Barroso E, Neff GW, Ranjan D, Toselli LT, Gane EJ, Scarola J, Alberts RG, Maller ES, Lo CM; Sirolimus Liver Conversion Trial Study Group. Sirolimus conversion regimen versus continued calcineurin inhibitors in liver allograft recipients: a randomized trial. Am J Transplant. 2012 Mar;12(3):694-705. doi: 10.1111/j.1600-6143.2011.03919.x. Epub 2012 Jan 10. PMID 22233522
- [Result] Backman L, Nicar M, Levy M, Distant D, Eisenstein C, Renard T, Goldstein R, Husberg B, Gonwa TA, Klintmalm G. FK506 trough levels in whole blood and plasma in liver transplant recipients. Correlation with clinical events and side effects. Transplantation. 1994 Feb 27;57(4):519-25. PMID 7509516
- [Result] Kong Y, Wang D, Shang Y, Liang W, Ling X, Guo Z, He X. Calcineurin-inhibitor minimization in liver transplant patients with calcineurin-inhibitor-related renal dysfunction: a meta-analysis. PLoS One. 2011;6(9):e24387. doi: 10.1371/journal.pone.0024387. Epub 2011 Sep 9. PMID 21931704
- [Result] Langone A, Steinberg SM, Gedaly R, Chan LK, Shah T, Sethi KD, Nigro V, Morgan JC; STRATO Investigators. Switching STudy of Kidney TRansplant PAtients with Tremor to LCP-TacrO (STRATO): an open-label, multicenter, prospective phase 3b study. Clin Transplant. 2015 Sep;29(9):796-805. doi: 10.1111/ctr.12581. Epub 2015 Aug 6. PMID 26113208
- [Result] Yoo MC, Vanatta JM, Modanlou KA, Campos L, Nezakatgoo N, Nair S, Eason JD. Steroid-free Liver Transplantation Using Rabbit Antithymocyte Globulin Induction in 500 Consecutive Patients. Transplantation. 2015 Jun;99(6):1231-5. doi: 10.1097/TP.0000000000000477. PMID 25539464
- [Result] Garnock-Jones KP. Tacrolimus prolonged release (Envarsus(R)): a review of its use in kidney and liver transplant recipients. Drugs. 2015 Feb;75(3):309-20. doi: 10.1007/s40265-015-0349-2. PMID 25613762
- [Result] Niel OR, Berthoux F, Albano L, Dahan P, Aoudia R, Gugenheim J, Cassuto E. Long-term glomerular filtration rate in liver allograft recipients according to the type of calcineurin inhibitors. Transplant Proc. 2009 Oct;41(8):3329-32. doi: 10.1016/j.transproceed.2009.09.034. PMID 19857743